CLINICAL TRIAL: NCT03108846
Title: Escitalopram for Agitation in Alzheimer's Disease
Acronym: S-CitAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dave Shade, Director, S-CitAD Coordinating Center, JHSPH Center for Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-CitAD; R01AG052510 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Dementia
Keywords: Alzheimer's Disease; Agitation
MeSH Terms: conditions — Dementia; Alzheimer Disease; Psychomotor Agitation | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Over-encapsulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Escitalopram (Experimental): Escitalopram up to 15mg/day taken as 1-3 capsules each containing 5mg escitalopram once per day in the morning
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): 1-3 capsules each containing placebo only once per day in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 5-15 mg/day (target: 15mg/day if tolerated)
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Masked placebo
  Other Names: non-applicable
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of escitalopram for agitation in Alzheimer's dementia.

DETAILED DESCRIPTION:
This study is designed to examine the efficacy and safety of escitalopram as treatment for agitation in Alzheimer's dementia (AD) patients. Participants with clinically significant agitation, and their caregiver(s), will receive a structured psychosocial intervention. Participants not showing a response three weeks later will be randomized 1:1 to escitalopram (up to 15 mg/day) or a matching placebo. Participants will receive study drug or placebo for 12 weeks, with in-person and remote (phone/video) visits at weeks 3, 6, 9, and 12, and with telephone contacts between in-person and remote visits. Participants who do show a response to the psychosocial intervention will not be randomized to study drug but will be followed remotely.

ELIGIBILITY:
Inclusion criteria

1. Alzheimer's dementia diagnosed clinically by the National Institute on Aging (NIA) and the Alzheimer's Association (AA) (2011 NIA/AA criteria)
2. Mini-Mental State Examination Telephone (MMSET) score of 3-20 inclusive
3. Meets the International Psychogeriatric Association (IPA) provisional criteria for agitation in cognitive disorders
4. Clinically significant agitation/aggression as assessed by the Neuropsychiatric Inventory (NPI) for which either:

   * The frequency is 'Very frequently,' or
   * The frequency is 'Frequently' AND the severity is 'Moderate' or 'Marked'
5. Provision of informed consent for participation in the study by both caregiver and participant (or, if participant is unable to provide informed consent, with surrogate consent and participant assent)
6. Availability of a caregiver who spends at least several hours per week with the participant, supervises his/her care, is willing to accompany the participant to study visits, and is willing to participate in the study
7. Stable (for ≥ 7 days) dosing of antipsychotics for agitation or psychosis, if being used at all
8. A medication for agitation is appropriate, in the opinion of the study physician

Exclusion criteria

1. Has major depression, as indicated by major depressive episode (MDE) in the past 90 days (meeting the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria)
2. Presence of another brain disease that fully explains the dementia, (e.g., extensive brain vascular disease, Parkinson's disease, dementia with Lewy bodies, traumatic brain injury, or multiple sclerosis)
3. Residence in a skilled nursing or Long-Term Acute Care (LTAC) facility
4. Contraindication to treatment with escitalopram as determined by a study physician, such as recent (30 days) use of monoamine oxidase inhibitors (MAOIs) or potential participant is hypersensitive to escitalopram or citalopram or any inactive ingredients
5. Prior failed treatment attempt with citalopram or escitalopram for agitation after adequate trial, at minimally accepted dose
6. Indication for psychiatric hospitalization or acute suicidality, in the opinion of the study physician
7. Recent (< 7 days) changes in antipsychotics, anticonvulsants, or psychosis (delusions or hallucinations) requiring a new or change in antipsychotic treatment (in the opinion of the study physician)
8. Abnormal corrected QT interval using Bazett's formula (QTcB)** as determined on enrollment ECG (defined as > 450 ms for men and > 470 ms for women)
9. Recent (30 days) presence of severely reduced renal function (as identified by a Glomerular filtration rate (GFR) clearance < 30 mL/min) or reduced hepatic function
10. Current treatment (within 7 days) with any of the following:

    * antidepressants (other than trazodone, ≤ 100 mg per day at bedtime)
    * benzodiazepines (other than lorazepam), or
    * psychostimulants
11. Recent (< 14 days) changes in Dextromethorphan/quinidine, prazosin, and pimavanserin
12. Recent (< 14 days) use of medical marijuana
13. Current participation in a clinical trial or in any study that may add a significant burden or affect neuropsychological or other study outcomes
14. Significant communicative impairments that would affect participation in a clinical trial
15. Any condition that, in the opinion of the study physician, makes it medically inappropriate or risky for the potential participant to enroll in the trial

    * if the QTcB is determined while the rhythm is paced, 50 ms is subtracted from the calculated value. The study cardiologist must confirm eligibility in this scenario.

Ages: 18 Years to 109 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
modified- Alzheimer's Disease Cooperative Study--Clinical Global Impression of Change (mADCS-CGIC) | after 12 weeks
  Clinical Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Lyketsos, MD, MHS, Study Chair — Johns Hopkins University
Locations (29):
- United States (22):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Biomedical Research Foundation, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Los Angeles/VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of Southern California Keck School of Medicine Memory and Aging Center, Los Angeles, California
  - Miami Jewish Health Systems, Miami, Florida
  - Kansas School of Medicine-Wichita Center for Clinical Research, Wichita, Kansas
  - Maryland VA Health Care System, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Bayview Medical Center, Baltimore, Maryland
  - Alzheimer Disease Center, Quincy, Massachusetts
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Abington Neurological Associates, Ltd, Abington, Pennsylvania
  - Alzheimer Disease Research Center; University of Pittsburgh, Pittsburgh, Pennsylvania
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Baylor AT&T Memory Center, Dallas, Texas
  - UT Health San Antonio, San Antonio, Texas
  - University of Virginia Adult Neurology, Charlottesville, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (7):
  - University of Calgary and Foothills Medical Centre, Calgary, Alberta
  - Lawson Health Research Institute/Parkwood Institute, London, Ontario
  - Neuropsychopharmacology Research Group, Sunnybrook, Toronto, Ontario
  - Unity Health, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Centre for Memory and Aging, Toronto, Ontario
  - Ontario Shores, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajji TK, Baksh SN, Shade DM, Ismail Z, Burhan AM, Okhravi HR, Padala PR, Rosenberg PB, Schneider LS, Porsteinsson AP, Lyketsos CG; S-CitAD Research Group. Escitalopram for agitation in Alzheimer's dementia: a randomized controlled phase 3 trial. Nat Med. 2025 May;31(5):1586-1591. doi: 10.1038/s41591-025-03569-y. Epub 2025 Mar 25. PMID 40133524
- [Derived] Ehrhardt S, Porsteinsson AP, Munro CA, Rosenberg PB, Pollock BG, Devanand DP, Mintzer J, Rajji TK, Ismail Z, Schneider LS, Baksh SN, Drye LT, Avramopoulos D, Shade DM, Lyketsos CG; S-CitAD Research Group. Escitalopram for agitation in Alzheimer's disease (S-CitAD): Methods and design of an investigator-initiated, randomized, controlled, multicenter clinical trial. Alzheimers Dement. 2019 Nov;15(11):1427-1436. doi: 10.1016/j.jalz.2019.06.4946. Epub 2019 Oct 3. PMID 31587995